CLINICAL TRIAL: NCT02830139
Title: A Phase II Study of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in the Treatment of Locally Advanced Colorectal Cancer During Radical Colorectal Resection
Brief Title: Radical Colorectal Resection and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Locally Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Bin Xiong, MD, Cancer Center of Wuhan University, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuhanU_HIPEC_colon
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Malignant Neoplasm of Colorectum
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy; Oxaliplatin; Capecitabine; Saline Solution; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radical colorectal resection without HIPEC (Sham Comparator): Patients will be treated with a radical colorectal resection for locally advanced colorectal cancer and postoperative chemotherapy (XELOX)
  Interventions: Procedure: Radical colorectal resection; Drug: Oxaliplatin , Capecitabine; Drug: Normal saline , Cisplatin , 5-Fu
- Radical colorectal resection with HIPEC (Experimental): Patients will be treated with a radical colorectal resection for locally advanced colorectal cancer and HIPEC with paclitaxel and 5-Fu and postoperative chemotherapy (XELOX)
  Interventions: Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC); Procedure: Radical colorectal resection; Drug: Oxaliplatin , Capecitabine

INTERVENTIONS:
Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) — Normal saline 3000ml-4000ml, Cisplatin 60mg/m2, 5-Fu 1500mg/m2, 43°C, 60min, During surgery and 7 days after surgery.
  Arms: Radical colorectal resection with HIPEC
Procedure: Radical colorectal resection — radical colorectal resection with lymphadenectomy
Drug: Oxaliplatin , Capecitabine — XELOX postoperative chemotherapy Oxaliplatin 130mg/m2 d1, Capecitabine 1000mg/m2 d1-14.
Drug: Normal saline , Cisplatin , 5-Fu
  Arms: Radical colorectal resection without HIPEC

SUMMARY:
The efficacy of HIPEC in prevention of local recurrence, distant metastasis or peritoneal metastasis in locally advanced colorectal cancer is not definite. The hypothesis of the trial is that radical colorectal resection plus HIPEC is superior to only radical colorectal resection in terms of overall survival.

DETAILED DESCRIPTION:
To determine the efficacy of HIPEC in the treatment of locally advanced colorectal cancer, patients are randomized into HIPEC group and control group. In HIPEC group, the patients undergo radical colorectal resection with lymphadenectomy and HIPEC with paclitaxel and 5-Fu. Patients in the control group just undergo radical colorectal resection with lymphadenectomy. Patients in both groups receive 8 cycles of postoperative chemotherapy (XELOX) and are followed up for 5 years or until death.

The trial is designed as a prospective, randomized, open, multicenter and parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Histological proved diagnosis of locally advanced colorectal cancer.
* No evidence of distant metastases or peritoneal metastases.
* Preoperative examination (CT/MRI) demonstrated resectable colorectal cancer with T3-T4 stage.
* Eligible for radical colorectal resection with lymphadenectomy.
* Have not received cytotoxic chemotherapy or radiotherapy.
* Written informed consent is obtained prior to commencement of trial treatment.

Exclusion Criteria:

* Existence of distant metastasis or peritoneal metastasis during surgery (M1).
* Any previous chemotherapy or radiotherapy
* Active systemic infections
* Inadequate cardiac function, renal function, liver function or bone marrow function at the beginning of the trial.
* Female patients who are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  From the date of surgery to the date of death or to the end of follow-up

SECONDARY OUTCOMES:
progression-free survival | 5 years
distant metastasis rate | 5 years
peritoneal metastasis rate | 5 years
local recurrence rate | 5 years
complication rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China